CLINICAL TRIAL: NCT01614769
Title: A Study to Assess the Effects of Glimepiride on Recovery From Hypoglycemia in Participants With Type 2 Diabetes Mellitus
Brief Title: Effects of Glimepiride on Recovery From Hypoglycemia in Participants With Type 2 Diabetes Mellitus (MK-0000-253)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-253
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo → Glimepiride 2 mg → Glimepiride 4 mg (Experimental): Participants received placebo in the first period, 2 mg glimepiride in the second period and 4 mg glimepiride in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp
- Glimepiride 2 mg → Glimepiride 4 mg → Placebo (Experimental): Participants received 2 mg glimepiride in the first period, 4 mg glimepiride in the second period and placebo in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp
- Glimepiride 4 mg → Placebo → Glimepiride 2 mg (Experimental): Participants received 4 mg glimepiride in the first period, placebo in the second period and 2 mg glimepiride in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp
- Placebo → Glimepiride 4 mg → Glimepiride 2 mg (Experimental): Participants received placebo in the first period, 4 mg glimepiride in the second period and 2 mg glimepiride in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp
- Glimepiride 2 mg → Placebo → Glimepiride 4 mg (Experimental): Participants received 2 mg glimepiride in the first period, placebo in the second period and 4 mg glimepiride in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp
- Glimepiride 4 mg → Glimepiride 2 mg → Placebo (Experimental): Participants received 4 mg glimepiride in the first period, 2 mg glimepiride in the second period and placebo in the third period, with a 7-day washout between each period.
  Interventions: Drug: Placebo; Drug: Glimepiride 2 mg; Drug: Glimepiride 4 mg; Procedure: Hypoglycemic Clamp

INTERVENTIONS:
Drug: Placebo — Two gross-matched glimepiride placebo tablets taken on Day -1 and Day 1 of the three treatment periods.
Drug: Glimepiride 2 mg — One placebo tablet and one 2-mg glimepiride tablet taken on Day -1 and Day 1 of the three treatment periods.
Drug: Glimepiride 4 mg — Two 2-mg glimepiride tablets taken on Day -1 and Day 1 of the three treatment periods.
Procedure: Hypoglycemic Clamp — On Day 1 of the three treatment periods, 180 minutes after drug treatment, a fixed-rate insulin infusion is combined with a variable-rate dextrose infusion to maintain plasma glucose concentrations at close to 50 mg/dL for 30 minutes.

SUMMARY:
This study aims to assess how glimepiride affects the recovery from hypoglycemia in participants with type 2 diabetes mellitus. The primary objective is to estimate the time taken by participants to recover from hypoglycemia to euglycemia after treatment with either 2 mg or 4 mg of glimepiride when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has clinically confirmed diagnosis of type 2 diabetes mellitus (T2DM) controlled by diet and exercise alone, or treated by metformin only with same dose for >= 12 weeks prior to screening visit.
* Females of reproductive potential who demonstrate nongravid state, agree to use (and/or have partner use) two acceptable methods of birth control starting at least two weeks prior to study, throughout study, and at least two weeks after last dose of study drug.
* Females of non-reproductive potential, post menopausal, status post hysterectomy, oophorectomy or tubal ligation.
* Is in good health, other than T2DM.
* Has been a nonsmoker and/or non user of nicotine-containing products for the previous 6 months. If discontinued use for previous 3 months, may be enrolled at investigator's discretion.
* Will follow American Heart Association weight maintaining diet and exercise program or equivalent beginning 2 weeks prior to study until poststudy visit.
* At screening visit has a Body Mass Index (BMI) =< 40 kg/m^2.
* At screening visit has a Hemoglobin A1c (HbA1c) of >= 7% and < 10% (+/- 0.1%).
* On the morning of randomization at predose has fasting plasma glucose (FPG) >= 126 mg/dL, and =< 250 mg/dL.

Exclusion Criteria:

* Has a history of stroke, chronic seizures, or major neurological disorder.
* Has a history of any illness that might confound the results of the study or pose additional risk to the participant.
* Has a history of type 1 diabetes mellitus, ketoacidosis, C-peptide =< 0.8 ng/mL, secondary forms of diabetes or diabetic complications.
* Has a history of neoplastic disease.
* Is a nursing mother.
* Has been treated =< one year of screening visit with sulfonylurea agents, meglitinides, dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) analogs, or insulin.
* Has received treatment within =< 12 weeks of screening visit with a peroxisome proliferator-activated receptor γ (PPARγ) agonist.
* Is taking medications for a co-morbid condition or anticipates taking new medications beginning 2 weeks prior to study.
* Consumes excessive amounts of alcohol or caffeinated beverages.
* Is a regular user of illicit drugs, or has a history of drug abuse within the previous 6 months.
* Has had major surgery, lost 500 mL of blood, or participated in another investigational study within 4 weeks prior to screening visit.
* Is on a weight loss program, but not in the maintenance phase, or treated with a weight loss medication within 8 weeks of prestudy visit.
* Has a history of severe allergies, anaphylactic reaction or intolerability to drugs, food, insulin, glimepiride or sulfonamide derivatives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07-18 (Actual); Primary Completion 2013-01-09 (Actual); Study Completion 2013-01-23 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Snyposis Link — http://www.merck.com/clinical-trials/study.html?id=0000-253&kw=0000-253&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Placebo → Glimepiride 2 mg → Glimepiride 4 mg | Glimepiride 2 mg → Glimepiride 4 mg → Placebo | Glimepiride 4 mg → Placebo → Glimepiride 2 mg | Placebo → Glimepiride 4 mg → Glimepiride 2 mg | Glimepiride 2 mg → Placebo → Glimepiride 4 mg | Glimepiride 4 mg → Glimepiride 2 mg → Placebo
Started | 2 | 1 | 2 | 2 | 1 | 2
Completed | 1 | 1 | 2 | 0 | 1 | 1
Not Completed | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Discontinued due to Hypoglycemia | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: 7-Day Washout
Arm/Group | Placebo → Glimepiride 2 mg → Glimepiride 4 mg | Glimepiride 2 mg → Glimepiride 4 mg → Placebo | Glimepiride 4 mg → Placebo → Glimepiride 2 mg | Placebo → Glimepiride 4 mg → Glimepiride 2 mg | Glimepiride 2 mg → Placebo → Glimepiride 4 mg | Glimepiride 4 mg → Glimepiride 2 mg → Placebo
Started | 1 | 1 | 2 | 0 | 1 | 1
Completed | 1 | 1 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo → Glimepiride 2 mg → Glimepiride 4 mg | Glimepiride 2 mg → Glimepiride 4 mg → Placebo | Glimepiride 4 mg → Placebo → Glimepiride 2 mg | Placebo → Glimepiride 4 mg → Glimepiride 2 mg | Glimepiride 2 mg → Placebo → Glimepiride 4 mg | Glimepiride 4 mg → Glimepiride 2 mg → Placebo
Started | 1 | 1 | 2 | 0 | 1 | 1
Completed | 1 | 1 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 7-Day Washout
Arm/Group | Placebo → Glimepiride 2 mg → Glimepiride 4 mg | Glimepiride 2 mg → Glimepiride 4 mg → Placebo | Glimepiride 4 mg → Placebo → Glimepiride 2 mg | Placebo → Glimepiride 4 mg → Glimepiride 2 mg | Glimepiride 2 mg → Placebo → Glimepiride 4 mg | Glimepiride 4 mg → Glimepiride 2 mg → Placebo
Started | 1 | 1 | 2 | 0 | 1 | 1
Completed | 1 | 1 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Placebo → Glimepiride 2 mg → Glimepiride 4 mg | Glimepiride 2 mg → Glimepiride 4 mg → Placebo | Glimepiride 4 mg → Placebo → Glimepiride 2 mg | Placebo → Glimepiride 4 mg → Glimepiride 2 mg | Glimepiride 2 mg → Placebo → Glimepiride 4 mg | Glimepiride 4 mg → Glimepiride 2 mg → Placebo
Started | 1 | 1 | 2 | 0 | 1 | 1
Completed | 1 | 1 | 1 | 0 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time From Hypoglycemia to Euglycemia
Description: Immediately after release of the hypoglycemic clamp, which maintained blood glucose close to 50 mg/dL, the time taken until glucose reached euglycemia, defined as 3 consecutive measurements >= 70 mg/dL, is called the recovery time.
Time Frame: From 1 to 180 minutes post hypoglycemic clamp
Population: The per-protocol population consisting of participants who received drug and completed the necessary post treatment measurements for at least one treatment period.
Measure: Least Squares Mean (90% Confidence Interval); unit: Minutes
Groups:
- Placebo: Participants received placebo in a treatment period.
- Glimepiride 2 mg: Participants received 2 mg Glimepiride in a treatment period.
- Glimepiride 4 mg: Participants received 4 mg Glimepiride in a treatment period.
Arm/Group | Placebo | Glimepiride 2 mg | Glimepiride 4 mg
Number analyzed (Participants) | 6 | 5 | 6
Minutes | 74.49 [48.20 to 100.77] | 88.90 [57.65 to 120.14] | 109.81 [81.05 to 138.57]
Statistical Analysis 1: Comparison: Placebo vs Glimepiride 2 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 14.41, 90% CI 2-sided [-22.98 to 51.80]
Statistical Analysis 2: Comparison: Placebo vs Glimepiride 4 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 35.33, 90% CI 2-sided [-2.08 to 72.74]

2. Primary Outcome: Rate of Recovery From Hypoglycemia to Euglycemia
Description: The rate of recovery is the difference in concentration between blood glucose at euglycemia and at the end of the hypoglycemic clamp, divided by the recovery time.
Time Frame: From 1 to 180 minutes post hypoglycemic clamp
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL/minute
Arm/Group | Placebo | Glimepiride 2 mg | Glimepiride 4 mg
Number analyzed (Participants) | 6 | 5 | 6
mg/dL/minute | 0.32 [0.24 to 0.40] | 0.22 [0.12 to 0.31] | 0.19 [0.10 to 0.27]
Statistical Analysis 1: Comparison: Placebo vs Glimepiride 2 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.10, 90% CI 2-sided [-0.21 to 0.00]
Statistical Analysis 2: Comparison: Placebo vs Glimepiride 4 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-0.24 to -0.03]

3. Primary Outcome: Incremental Weighted Average Blood Glucose Concentration Over 3 Hours of Hypoglycemic Recovery
Description: The incremental weighted average qualitatively assesses overall hypoglycemic recovery by measuring mean glycemia over the 3 hour recovery period. Blood glucose measured at the release of the hypoglycemic clamp, considered the baseline value, was subtracted from blood glucose values measured over the ensuing 3 hours of hypoglycemic recovery. These differences from baseline were averaged to calculate the incremental weighted average blood glucose concentration.
Time Frame: From 1 to 180 minutes post hypoglycemic clamp
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Glimepiride 2 mg | Glimepiride 4 mg
Number analyzed (Participants) | 6 | 5 | 6
mg/dL | 22.61 [17.55 to 27.68] | 17.58 [11.78 to 23.38] | 15.34 [9.94 to 20.75]
Statistical Analysis 1: Comparison: Placebo vs Glimepiride 2 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -5.03, 90% CI 2-sided [-11.12 to 1.05]
Statistical Analysis 2: Comparison: Placebo vs Glimepiride 4 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -7.27, 90% CI 2-sided [-13.30 to -1.24]

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug
Arm/Group | Placebo | Glimepiride 2 mg | Glimepiride 4 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/9 | 2/6 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Glimepiride 2 mg (N=6) | Glimepiride 4 mg (N=7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.